CLINICAL TRIAL: NCT00842348
Title: Open Label Extension Study of Lanreotide Autogel 120 mg in Patients With Non-functioning Entero-pancreatic Endocrine Tumour
Brief Title: Study of Lanreotide Autogel 120 mg in Patients With Non-functioning Entero- Pancreatic Endocrine Tumour
Acronym: NET729
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-55-52030-729; 2008-004019-36 (EudraCT Number)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Non Functioning Entero-pancreatic Endocrine Tumour
Keywords: Lanreotide; Somatuline; Neuroendocrine tumour; NET
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lanreotide (Autogel formulation) (Experimental): Patients from the preceding DB study (Study 726) were treated with open label lanreotide Autogel 120 mg by deep subcutaneous injections every 28 days. Patients were included if they had been treated with lanreotide (Autogel formulation) or placebo in DB Study 726 and had stable disease at the end of the 96-week treatment period, or if they had received placebo and had disease progression at any time during Study 726. Safety data were based on the safety population patients who received lanreotide in Study 729). The main efficacy analysis was based on the ITT population (patients randomised in Study 726 regardless of whether they continued into Study 729).
  Interventions: Drug: lanreotide (Autogel formulation)

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — Autogel 120 mg
  Other Names: Lanreotide; Lanreotide Autogel; Somatuline; Somatuline Autogel; Somatuline Depot

SUMMARY:
The primary purpose of this extension study was to assess the long term safety of patients with nonfunctioning enteropancreatic neuroendocrine tumour (NET), who were treated with open label lanreotide Autogel (120 mg every 28 days) and who participated in a previous study, 2-55-52030-726 (NCT00353496).

DETAILED DESCRIPTION:
While somatostatin analogue treatment is the primary medical therapy for patients with hormone related symptoms and is indicated for the treatment of hormone related symptoms in many international countries, there is no reference standard medical therapy for asymptomatic patients. A 96-week study (Study 2-55-52030-726 (726), NCT00353496) was conducted to investigate the effect of lanreotide Autogel on progression free survival (PFS) in patients with well or moderately differentiated nonfunctioning enteropancreatic NET. While Study 726 was ongoing, the sponsor considered that therapy with lanreotide Autogel should continue to be an option to patients with stable disease at the end of the 96-week treatment period. This extension study was therefore initiated (Study 2-55-52030-729 (729)) which investigated the long term safety of treatment with lanreotide Autogel and enabled investigators to continue to treat their patients who had stable disease, as well as to treat placebo patients who experienced disease progression during the initial 96-week study (Study 726).

ELIGIBILITY:
Inclusion Criteria:

1. Had provided written informed consent prior to any study-related procedures.
2. Had been enrolled and treated in Study 2-55-52030-726 and either:

   * Was stable at 96 weeks of treatment (whatever the treatment received during the 2 years of participation, i.e. no code break at Week 96); or,
   * Had received at least one injection in Study 2-55-52030-726 and had disease progression, confirmed by central assessment, during the course of the study and code break showed placebo.
3. Had a World Health Organisation (WHO) performance score lower than or equal to 2.

Exclusion Criteria:

1. Had been enrolled and treated in the frame of the protocol and had disease progression during the study and the code break showed a treatment with lanreotide Autogel 120 mg.
2. Had received any new treatment for the entero-pancreatic NET since the end of participation in the study.
3. Were likely to require any additional concomitant treatment to lanreotide Autogel 120 mg for the entero-pancreatic NET.
4. Had been treated with radionuclide at any time prior to study entry.
5. Had a history of hypersensitivity to drugs with a similar chemical structure to lanreotide Autogel 120 mg.
6. Were likely to require treatment during the study with drugs that were not permitted by the study protocol.
7. Were at risk of pregnancy or lactation. Females of childbearing potential had to provide a negative pregnancy test at the start of study and had to be using oral, double barrier or injectable contraception. Non-childbearing potential was defined as postmenopause for at least 1 year, or surgical sterilisation or hysterectomy at least 3 months before the start of the study.
8. Had any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
9. Had abnormal findings at Visit 1, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might have jeopardised the patient's safety or decreased the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.
10. Previous enrolment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (25):
- United States (2):
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - The Johns Hopkins Hospital, Baltimore, Maryland
- Belgium (2):
  - UZ Antwerpen, Antwerp
  - UCL Saint Luc, Brussels
- Czechia (2):
  - Fakultni nemocnice Na Bulovce, Prague
  - General faculty, Prague
- France (4):
  - Hôpital Beaujon, Clichy
  - CAC Oscar Lambret, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hôpital R. Debré, Reims
- Italy (4):
  - Centro di Refierimiento Oncologica, Aviano
  - INSCT, Milan
  - University of Naples, Naples
  - Azienda San Giovanni Battista, Torino
- Poland (2):
  - Centrum Diagnostyczno-Lecznicze "Gammed", Warsaw
  - Zaklad Diagnosttyki Radiologicznej, Centralny Szpital Klincny, Warsaw
- Narodny onkologicky ustav, Bratislava, Slovakia
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Institut Catala Oncologia, Barcelona
- United Kingdom (6):
  - University Hospital Wales, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James Hospital, Leeds
  - Royal Free Hospital, London
  - QMC, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Gomez-Panzani E, Ruszniewski P; CLARINET Investigators. Anti-tumour effects of lanreotide for pancreatic and intestinal neuroendocrine tumours: the CLARINET open-label extension study. Endocr Relat Cancer. 2016 Mar;23(3):191-9. doi: 10.1530/ERC-15-0490. Epub 2016 Jan 7. PMID 26743120
- [Derived] Caplin ME, Pavel M, Phan AT, Cwikla JB, Sedlackova E, Thanh XT, Wolin EM, Ruszniewski P; CLARINET Investigators. Lanreotide autogel/depot in advanced enteropancreatic neuroendocrine tumours: final results of the CLARINET open-label extension study. Endocrine. 2021 Feb;71(2):502-513. doi: 10.1007/s12020-020-02475-2. Epub 2020 Oct 14. PMID 33052555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 26 active sites across 10 countries in Study 729; however, only 24 recruited patients. The study was initiated in February 2009 and was completed in December 2015.
Groups:
- Lanreotide Autogel: Patients who received lanreotide 120 mg (Autogel formulation) in the preceding double blind (DB) study (Study 2-55-52030-726) and who continued to receive lanreotide 120 mg (Autogel formulation) in the open label study.
- Placebo: Patients who received placebo in the preceding DB study (Study 2-55-52030-726) and who received lanreotide 120 mg (Autogel formulation) in the open label study.
Period: Patients Randomised in Study 726
Arm/Group | Lanreotide Autogel | Placebo
Started | 101 | 103
Completed | 42 (41 patients had stable disease and 1 patient had progressive disease.) | 47 (15 patients had stable disease and 32 patients had progressive disease.)
Not Completed | 59 | 56
Not completed — Did not enter Study 729 | 59 | 56
Period: Study 729
Arm/Group | Lanreotide Autogel | Placebo
Started | 42 | 47
Completed | 16 (Enrolled in Study 729 and received at least one dose of open label lanreotide Autogel.) | 9 (Enrolled in Study 729 and received at least one dose of open label lanreotide Autogel.)
Not Completed | 26 | 38
Not completed — Disease progression/death | 19 | 30
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Due to Sponsor stopping the study | 1 | 1
Not completed — Due to non-availability of IP | 0 | 1
Not completed — Sponsor's decision | 1 | 0
Not completed — Surgical resection | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients who received at least one dose of lanreotide Autogel in Study 729.
Groups:
- Lanreotide Autogel: Patients who received lanreotide 120 mg (Autogel formulation) in the preceding DB study (Study 2-55-52030-726) and who continued to receive lanreotide 120 mg (Autogel formulation) in the open label study.
- Total: Total of all reporting groups
Arm/Group | Lanreotide Autogel | Placebo | Total
Number analyzed (Participants) | 42 | 47 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.8) | 61.3 (10.2) | 62.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 19 | 25 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 3 | 3
  Black or African American | 1 | 0 | 1
  Caucasian/White | 41 | 44 | 85

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Adverse events (AEs) that were ongoing from Study 726 at the time of entry into Study 729 were transcribed into the case report form (CRF) for Study 729 with a start date corresponding to the original report of this AE in Study 726. All new AEs that started after the last visit in Study 726 (i.e. irrespective of whether the AE had onset before or after giving informed consent for Study 729) were recorded Study 729.
  An AE was considered as a treatment emergent adverse event (TEAE) for Study 729 if:
  * It was not present prior to receiving the first dose of study treatment in Study 729; or,
  * It was present prior to receiving the first dose of study treatment in Study 729 but the intensity increased after the first dose of study treatment in Study 729.
  Adverse event data are presented in the AE section.
Time Frame: Throughout the study until the completion/early discontinuation visit.
Population: Safety population: all patients who received at least one dose of lanreotide Autogel in Study 729.
Measure: Number; unit: participants with any TEAEs
Groups:
- Placebo: Patients who received placebo in the preceding double DB study (Study 2-55-52030-726) and who received lanreotide 120 mg (Autogel formulation) in the open label study.
- Total: All patients treated with Lanreotide 120 mg (Autogel formulation) in the open label study.
Arm/Group | Lanreotide Autogel | Placebo | Total
Number analyzed (Participants) | 42 | 47 | 89
participants with any TEAEs | 40 | 46 | 86

2. Secondary Outcome: Progression Free Survival (PFS): Kaplan-Meier Estimate
Description: The time from randomisation in Study 726 to the first occurrence of either disease progression (measured using Response Evaluation Criteria In Solid Tumours [RECIST] criteria) or death in Study 726 or in Study 729, or equivalently, the Progression Free Survival (PFS) time.
  Tumour assessments for the placebo group after switching to open label lanreotide Autogel were excluded for the purpose of this analysis. Estimation of the median was based on the Kaplan-Meier method.
Time Frame: Throughout the study (every 24 weeks and at completion/withdrawal visit)
Population: Intention-to-treat (ITT) population: all patients randomised in the original protocol Study 726 (regardless of whether they continued into the extension Study 729). The ITT population was analysed using patients as randomised in Study 726.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Lanreotide Autogel - Randomised Treatment in Study 726: All patients randomised to lanreotide 120 mg (Autogel formulation) in the original protocol Study 726 (regardless of whether they continued into the extension Study 729).
- Placebo - Randomised Treatment in Study 726: All patients randomised to placebo in the original protocol Study 726 (regardless of whether they continued into the extension Study 729).
Arm/Group | Lanreotide Autogel - Randomised Treatment in Study 726 | Placebo - Randomised Treatment in Study 726
Number analyzed (Participants) | 101 | 103
weeks | 154.14 [123.57 to 237.43] | 72.00 [48.43 to 84.57]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time that the patient withdrew or completed Study 726 until withdrawal in Study 729.
Description: Adverse events were elicited by direct, nonleading questioning or by spontaneous reports. Local tolerance AEs were assessed by spontaneous reports. Any local tolerance assessed as present and judged as clinically significant was recorded as an AE in the CRF. Pre-existing conditions that worsened during the study were reported as AEs. Adverse events that were ongoing at the end of Study 726 were recorded and followed during Study 729.
Arm/Group | Lanreotide Autogel | Placebo | Total
Serious Adverse Events (participants affected / at risk) | 11/42 | 14/47 | 25/89
Other Adverse Events (participants affected / at risk) | 34/42 | 42/47 | 76/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (N=42) | Placebo (N=47) | Total (N=89)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (2)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (N=42) | Placebo (N=47) | Total (N=89)
Diarrhoea (Gastrointestinal disorders) | 8 (28) | 15 (25) | 23 (53)
Nausea (Gastrointestinal disorders) | 7 (15) | 6 (11) | 13 (26)
Constipation (Gastrointestinal disorders) | 5 (8) | 4 (6) | 9 (14)
Vomiting (Gastrointestinal disorders) | 7 (8) | 5 (11) | 12 (19)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (9) | 14 (16)
Abdominal discomfort (Gastrointestinal disorders) | 3 (5) | 2 (3) | 5 (8)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (4) | 7 (9)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 9 (9) | 12 (13)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 4 (7) | 7 (10)
Steatorrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 7 (7)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (12) | 10 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (10) | 9 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 3 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 3 (6) | 7 (7) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 1 (1) | 5 (7)
Viral infection (Infections and infestations) | 4 (5) | 2 (2) | 6 (7)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (6) | 7 (8)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (9) | 5 (10)
Dizziness (Nervous system disorders) | 4 (6) | 2 (2) | 6 (8)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 4 (5) | 8 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 4 (5)
Weight decreased (Investigations) | 1 (1) | 3 (5) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3) | 7 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 4 (6)
Fatigue (General disorders) | 5 (6) | 4 (6) | 9 (12)
Oedema peripheral (General disorders) | 3 (4) | 1 (1) | 4 (5)
Injection site pain (General disorders) | 1 (1) | 3 (3) | 4 (4)
Asthenia (General disorders) | 0 (0) | 4 (4) | 4 (4)
Injection site nodule (General disorders) | 0 (0) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 3 (5) | 3 (5)
Insomnia (Psychiatric disorders) | 4 (5) | 0 (0) | 4 (5)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 7 (10) | 7 (9) | 14 (19)
Hypertension (Vascular disorders) | 4 (4) | 5 (5) | 9 (9)
Flushing (Vascular disorders) | 1 (1) | 3 (5) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6) | 6 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 6 (7)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (6) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor required reasonable opportunity to review any abstract, presentation, or paper before the material is submitted for publication or communicated. This also applied to any amendments that are requested by referees or journal editors. The Sponsor committed to comment on the draft documents within a time period agreed in the contractual arrangements between the Sponsor and authors or their institution. Delays were also possible if publication would adversely affect patentability.